CLINICAL TRIAL: NCT04200040
Title: A Phase II Clinical Study to Evaluate the Safety and Efficacy of OrienX010 in Previously Untreated With Dacarbazine Patients in Unresectable Stage IIIb/IIIc or Stage IV(Mla/Mlb) Malignant Melanoma
Brief Title: A Clinical Study to Evaluate the Safety and Efficacy of OrienX010 in Unresectable Malignant Melanoma Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: OrienGene Biotechnology Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OrienX010-II-21
Record Dates: First submitted 2019-12-10; First posted 2019-12-16 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Melanoma (Skin)
MeSH Terms: conditions — Melanoma | interventions — Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): OrienX010 will be administered once every two weeks by intratumoral injection. The treatment dose , depends on the patient's tumour size, The maximum dose of OrienX010 in at each treatment , the expected accumulated dose in 10 mL. The investigator should be confirmed the injectable tumor size and adequate dose within 24 hours prior to treatment.
  OrienX010 treatment will be continuous and extend from first dose of study medication until to complete response, clinical related progression disease (PDr), untolerated toxicities, lost to follow up, death or meet end of treatment criteria.
  Interventions: Biological: OrienX010 injection
- Control group (Active Comparator): Dacarbazine will be administered once every three weeks by intravenous 1000mg/square meter. Dacarbazine treatment will be continuous and extend from first dose of study medication until to progression disease (PD), untolerated toxicities, lost to follow up, death or meet end of treatment criteria.
  Interventions: Drug: Dacarbazine (DTIC)

INTERVENTIONS:
Biological: OrienX010 injection — OrienX010 to be used in this study have been developed and manufactured by OrienGene Biotechnology Ltd.
  Dacarbazine to be used in this study was manufactured by Sinopharm A-Think Pharmaceutical Co., Ltd.
  Other Names: Recombinant Human GM-CSF Herpes Simplex Virus Injection
  Arms: treatment group
Drug: Dacarbazine (DTIC) — Dacarbazine to be used in this study was manufactured by Sinopharm A-Think Pharmaceutical Co., Ltd.
  Arms: Control group

SUMMARY:
This study is being performed to evaluate the safety and efficacy of Dacarbazine and OrienX010 therapy in Untreated Patients With Unresectable Stage IIIb/IIIc or Stage IV(Mla/Mlb) Melanoma.

The study will be conducted in about 6 centres in China and total 165 patients will be enrolled. All eligible Patients will be randomized between Dacarbazine and OrienX010 in a 1:2 ratio, so 1/3 (55) patients will receive the Dacarbazine and 2/3 (110) patients will receive the OrienX010.

During the treatment phase, the patient will receive OrienX010 administration once biweekly or Dacarbazine once every 3 week until to the end of treatment (EOT). The duration of safety follow-up for adverse events (AEs) and serious adverse events (SAEs) will be to 90 days after the end of treatment. The details please refer to study schema.

For patients who have completed the study treatment and no disease progression, follow-up visits will take place every 3 months after the end of treatment visit until the occurrence of disease progression. If disease progression occurred, the investigator will collect the anticancer treatment information and survival of individuals until 80% death event.

After the end of study, if patient want to continue receiving the OrienX010 treatment and judged by investigator, sponsor will provide OrienX010 and Dacarbazine for free until disease progression/death or OrienX010 on marketing launch.

ELIGIBILITY:
Inclusion Criteria:

1. Obtain the current IRB approved informed consent with written from potential patients before the any screening activities or procedures.
2. Male or female, ≥ 18 years and ≤ 70 years of age.
3. Patients with histologically proven unresectable stage IIIb /IIIc or IV (M1a/M1b) malignant melanoma following AJCC edition 8 published 2016 guidance. If patient in stage IV (M1b), pulmonary lesion as following:

   number of pulmonary lesion must be ≤ 5; any single lesion must less than 20 mm in longest diameter; total cumulative diameter of all lesions must be ≤ 50 mm;
4. Patients with at least one measurable lesion with size ≥ 10 mm and < 100mm.
5. Patient with at least one injectable lesion (long diameter ≥ 10 mm and < 100mm
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
7. Patients with life expectancy > 5 months as judged by investigator.
8. Patients with adequate bone marrow, liver and renal function within 28 days prior to study entry, as defined by the following:

   * White Blood Cell count ≥3.0 × 109/L
   * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
   * Platelet count≥ 100 × 109/L
   * Hemoglobin > 10.0 g/dl.
   * Albumin ≥ 3 g/dl.
   * liver function: Total bilirubin ≤ 1.5 x upper normal limit (UNL) , Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x upper normal limit (UNL).
   * renal function: serum creatinine < 1.5 x UNL or 24 hour creatinine clearance rate≥ 50 mL/min（calculated by Cockcroft and Gault）
   * International normalized ratio (INR) < 1.5 and Activated partial thromboplastin time (APTT) or Partial thromboplastin time (PTT) ≤ 1.5 × ULN
9. Subjects who have received any anti-cancer therapy, including radiotherapy, cytotoxic, hormonal, biological (including humanized antibodies) and targeted agents within 28 days, or five half-lives of the drug (whichever is longer) prior to randomization and not recovered from acute toxicities as a result of prior anti-cancer therapy to less than or equal to Grade 1, according to Common Terminology Criteria for Adverse Events (CTCAE, version 4.03).
10. Women of childbearing potential （early menopause, Post-menopause < 2 years and non- sterilization）, Man and man with female partner of childbearing potential should be use effective contraception during the study period , e.g. sterilization, progestogen oral contraceptives, injectable progestogen, implants of levonorgestrel, oestrogenic vaginal ring, percutaneous contraceptive patches or intrauterine device (IUD) or intrauterine system (IUS), abstinence or or double barrier method (condom or occlusive cap plus spermicidal agent).

Exclusion Criteria:

1. Patients that have previously been treated with dacarbazine.
2. Previous treatment with any investigational product or T-VEC or other similar ' oncolytic' viruses therapy.
3. Sizes of tumor does not meet the requirement of injection or unacceptable for intratumoral injection.
4. Patients who have treatment with anti-HSV antiviral therapy (such as acyclovir, ganciclovir, foscarnet, etc.) within 4 weeks prior to the first IP administration.
5. No history of malignancy within the past 5 years except for the following: adequately treated of stage I or II basal cell/squamous cell skin cancer, superficial bladder cancer or any other cancer from which the patient has been completed curative therapy.
6. Patients with known or suspected allergies and/or hypersensitivity to any component of OrienX10 or Dacarbazine.
7. HSV - 1 antibody IgG and IgM are negative
8. Positive test for hepatitis B virus surface antigen (HBVsAg) and HBV DNA copies >1x103copies /mL.
9. Positive test for hepatitis C and Human Immunodeficiency Virus (HIV) Patients with clinically evident Hepatitis C virus (HCV) and Human Immunodeficiency Virus (HIV) infection.
10. Patient with uncontrolled systemic illness including, but not limited to, serious infection, uncontrolled, diabetes, unstable angina, cerebrovascular accidents or transient ischaemic attack, myocardial infarction, congestive heart failure, clinically significant arrhythmias not controlled by medication, liver, kidney or metabolic disease.
11. Patient with autoimmune diseases.
12. Patient has psychological or psychiatric disorder or alcohol dependence or Drug addiction which would increase risk or limit compliance with study requirements or influence the study result.
13. Use of any investigational drugs, biologics, or devices within 30 days prior to screening visit or planned use during the course of study.
14. Pregnant or breastfeeding women or women desiring to become pregnant within the timeframe of the study or women/men of reproductive potential not using an effective contraception.
15. Any condition, judged by investigator, that shows subjects are not suitable for participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2017-08-27 (Actual); Primary Completion 2022-12-27 (Estimated); Study Completion 2022-12-27 (Estimated)

PRIMARY OUTCOMES:
PFS | Every 12 weeks until subjects disease progressive, an average of 24 weeks
  Progression-free survival (PFS), defined as the first documentation of objective disease progression, according to Response Evaluation Criteria in Solid Tumors (RECIST v.1.1)

SECONDARY OUTCOMES:
DCR | through study completion, an average of 1 year
  Disease Control Rate (DCR), defined as the proportion of subjects with complete response, partial response, or stable disease for more than 3 months, according to RECIST v.1.1 criteria
ORR | through study completion, an average of 1 year
  Objective Response Rate (ORR), defined as complete or partial tumor response, according to RECIST v.1.1 criteria
OS | Approximately 3 years
  Overall survival defined as the time from randomization to death from any cause
DRR | through study completion, an average of 1 year
  Durable response rate (DRR) defined as objective response lasting continuously ≥ 6 months
Quality of life assessment | every 6 weeks up to 24 weeks, and then every 12 weeks up to the date of end of treatment,an average of 24 weeks
  Use EORTC QLQ-C30 to assess quality of life. The EORTC(European Organization for Research and Treatment of Cancer) QLQ-C30 (Quality of Life Questionnaire C30), is a cancer-specific quality of life instrument applicable to a broad range of cancer patients.
  QLQ-C30 contain 15 domain, The standard score for each domain from 0-100. higher scores mean a worse outcome.
Incidence of treatment-related SAE and AE | From date of enrolling to 90 days after end of treatment
  Number of participants with treatment-related serious adverse events (SAE) and adverse events that assessed by CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No